CLINICAL TRIAL: NCT04033198
Title: Senior House Officer of Trauma and Emergency Surgery
Brief Title: Clinicopathological Aspects of Acute Appendicitis in Patients Above Age of Thirty at Sulaimani Emergency Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Maha Sabawi, Senior house officer of trauma and emergency surgery, University of Sulaimani
Other Study IDs: AA8
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Acute Appendicitis in Elderly
Keywords: Clinico-pathology , acute appendicitis , elderly , aging , histopathology
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- fourth decade: appendectomy done , appendix send for histopathological examination
  Interventions: Procedure: Appendectomy
- fifth decade: appendectomy done , appendix send for histopathological examination
  Interventions: Procedure: Appendectomy
- sixth decade: appendectomy done , appendix send for histopathological examination
  Interventions: Procedure: Appendectomy
- older than 60 years: appendectomy done , appendix send for histopathological examination
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — patients diagnosed as acute appendicitis , appendectomy done

SUMMARY:
Aims of this study are :

* Estimate the incidence of A.A. in patients above age of 30 y in 4 age groups .
* Correlate between different clinical aspects and histopathological results.
* Determine rate of negative appendectomy in those patients.

DETAILED DESCRIPTION:
Acute appendicitisis the clinical condition which refer to inflammation of the vermiform appendix1. It is the most common abdominal emergency2,3,4 .it accounts for more than 40,000 hospital admissions in England every year 5 . Approximately 8% of the population in Western countries would have appendicitis during their life 6 .In the United States, the estimated incidenc of acute appendicitis is 11 cases per 10,000 population 5 . However, in South Africa, the incidencewas estimated to be less than 9 per 100,000 6 .Appendectomy is considered the most common emergency surgical procedure worldwide6,8 ,9. The cause of acute appendicitis is unknown but it is multifactorial; luminal obstruction , dietary and familial factors have been suggested 5 . Fecoliths are the most common cause of obstruction. It was demonstrated that the mean duration of abdominal pain in patients with gangrenous appendix is 46.2 hours and 70.9 hs for perforated 7 .

The peak incidence of acute appendicitis is at the age of 10 to 30 years 6,10. There are special features for appendicitis according to age 1. A.A is primarily a disease of the younger population, with only 5-10% of cases occurring in elderly people, but the incidence of acute appendicitis in elderly began to increase with the increase in life expectancy14. Older patients with acute abdominal pain are high-risk patients, unlike their younger counterparts15 . Morbidity and mortality rates are greater in elderly due to atypical presentations and delay in diagnosis leading to increase rate of perforation and intra-abdominal infection.. They need to be clinically evaluated by experienced surgeons within a narrow time margin14,15.

ELIGIBILITY:
Inclusion Criteria:

* patients above age of thirty appendectomy done for them

Exclusion Criteria:

* patients less than thirty years conservative mangement

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes 70 patients with age above than thirty years old. The patients are divided into 4 age groups :group 1 (30-39 y) , group 2(40-49), group 3(50-59) and group4 (patients older than 60 y) .They were admitted to our emergency hospital with features of acute appendicitis. A detailed history was taken and clinical examination of the patient was carried out at the time of admission .Data was collected regarding investigations (CBC , GUE , US). Appendectomy done for the 70 patient,their operative findings along with any complications as well as histopathological findings were recorded
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Clinico -pathological aspects of acute appendicitis in patients above age of thirty in Sulaimani Emergency hospital | 2 month
  perform appendectomy for all the patients who diagnosed as acute appendicitis